CLINICAL TRIAL: NCT03092752
Title: Clinical Characteristics and Practice Patterns of Type 2 Diabetes Mellitus (T2D) Patients Treated With Oral Antidiabetic Drugs (OAD) in Japan: Analysis of Medical and Health Care Database of the Medical Data Vision (MDV)
Brief Title: Clinical Characteristics and Practice Patterns of Type 2 Diabetes Mellitus Patients Treated With OADs in Japan: Analysis of Medical and Health Care Database of the MDV
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1218.178
Record Dates: First submitted 2017-02-20; First posted 2017-03-28 (Actual); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Hypoglycemic Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Patients with T2DM
  Interventions: Drug: oral antidiabetic drugs

INTERVENTIONS:
Drug: oral antidiabetic drugs — OADs usage conditions and dose selection in T2DM patients

SUMMARY:
Appropriate use of oral antidiabetic drugs (OADs) including dose-reduction is important for patient's safety in T2DM patients with renal impairment (RI). However, there are insufficient data on dose adjustment in accordance with the prescription pattern and the risk of RI of OADs, in particular Dipeptidyl-peptidase-4 inhibitors, in clinical practice in Japan. Therefore, we will investigate OADs usage conditions and dose selection in T2DM patients with RI in clinical practice in Japan

ELIGIBILITY:
Inclusion criteria:

* Patients with T2DM (ICD code: E11 or E14).
* Patients must have their first prescription (defined as index date*) for any study drugs between 01/01/2014 and 30/09/2016.
* Patients must have at least 6 months enrolment verified by the presence of any record except for the study drug prescriptions within the database (look back period) prior to the index date for each drug.

Exclusion criteria:

* Patients who were under 40 years at the time of diagnosis of diabetes.
* Patients with record of type 1 diabetes mellitus.
* Patients who prescribed the study drugs during 6 month prior to index date for each drug.
* Patients whose mean visit interval are more than 92 days

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Japan
Sampling Method: Non-Probability Sample
Enrollment: 162116 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Medical Data Vision Co. Ltd, Shinagawa-ku, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a retrospective observational cohort study. The data was taken from Medical Data Vision (MDV) database for the duration from 1st January 2014 to 30th September 2016 .
Pre-assignment Details: The data of 523585 patients was available in the MDV database having a diagnosis of Type 2 Diabetes Mellitus (T2DM) of which data of 162116 eligible patients was included in this study.
Groups:
- Oral Antibiotic Drugs: Patients with type 2 diabetes mellitus (T2DM) were treated with oral antibiotic drugs (OAD) such as Dipeptidyl-peptidase 4 inhibitors, sulfonylureas, biguanides, thiazolidinediones, α-glucosidase and glinides as per prescription in Japan.
Period: Overall Study
Arm/Group | Oral Antibiotic Drugs
Started (Data for these patients was available in database.) | 523585
Completed (These many patients satisfies the inclusion criteria and hence included in the study.) | 162116
Not Completed | 361469
Not completed — Aged <40 years | 14209
Not completed — At least one claim with T2DM | 61299
Not completed — Having no claim of study drugs | 29282
Not completed — Average hospital visit interval >92 days | 10779
Not completed — <6 month history | 245900

BASELINE CHARACTERISTICS:
Population: Baseline data is presented for eligible T2DM patients for inclusion.
Arm/Group | Oral Antibiotic Drugs
Number analyzed (Participants) | 162116
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.7 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63055
  Male | 99061
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Secondary Outcome: Number of Prescriptions of OAD by Each Renal Impairment (RI) Stages
Description: This outcome observes number of index dates for each class of OAD as per RI classes. RI classes were defined based on eGFR values. Results observed were based on index dates used for comparing drugs between the classes.
Time Frame: Within 6 months from index date
Population: All index dates computed from patients with eGFR data, included in the study were considered for this analysis. Some patients were prescribed for more than one study drug and thus we can observe more number of index dates than number of patients.
Measure: Number; unit: Prescriptions
Groups:
- Group G1: The group 1 (G1) contains patients (prescribed for OADs) with renal function stage as normal. Normal renal function stage is defined based on serum creatinine value for males between 0.6 milligram per deciLitre and 1.2 milligram per deciLitre and that for females is between 0.4 milligram per deciLitre and 0.9 milligram per deciLitre.
- Group G2: The group 2 (G2) contains patients (prescribed for OADs) with renal function stage as mild. Mild renal function stage is defined based on serum creatinine value for males between 1.2 milligram per deciLitre and 1.4 milligram per deciLitre and that for females is between 0.9 milligram per deciLitre and 1.2 milligram per deciLitre.
- Group G3: The group 3 (G3) contains patients (prescribed for OADs) with renal function stage as moderate. Moderate renal function stage is defined based on serum creatinine value for males between 1.4 milligram per deciLitre and 2.4 milligram per deciLitre and that for females is between 1.2 milligram per deciLitre and 2.0 milligram per deciLitre.
- Group G4+: The group 4+ (G4+) contains patients (prescribed for OADs) with renal function stage as severe or end stage kidney disease (ESKD). Severe or ESKD renal function stage is defined based on serum creatinine value greater than 2.4 milligram per deciLitre for males and greater than 2.0 milligram per deciLitre for females.
- Total: Total for all participants
Arm/Group | Group G1 | Group G2 | Group G3 | Group G4+ | Total
Number analyzed (Participants) | 3868 | 11188 | 7776 | 2554 | 206406
Prescriptions
  DPP4 inhibitors | 1592 | 4877 | 3566 | 1411 | 11446
  Biguanides (BG) | 838 | 2373 | 1045 | 67 | 4323
  Sulfonylurea (SU) | 530 | 1446 | 1090 | 208 | 3274
  α-glucosidase (AGI) | 429 | 1175 | 1055 | 488 | 3147
  Glinide | 252 | 691 | 610 | 337 | 1890
  Thiazolidinedione (TZD) | 227 | 626 | 410 | 43 | 1306

2. Primary Outcome: Number of Index Dates
Description: The date at which patients having their first prescription for any study drugs between 1st January 2014 and 30th September 2016 is defined as index date. Results observed were based on index dates used for comparing drugs between the classes. The reported data represent the number of time a prescription was written between 1st January 2014 and 30th September 2016.
Time Frame: From 1st January 2014 to 30th September 2016 (At index date)
Population: All index dates computed from patients included in the study were considered for this analysis. Some patients were prescribed for more than one study drug and thus we can observe more number of index dates than number of patients.
Measure: Number; unit: Number of Prescriptions
Groups:
- Oral Antibiotic Drugs: Patients with type 2 diabetes mellitus (T2DM) were treated with oral antibiotic drugs (OAD) such as Dipeptidylpeptidase 4 inhibitors, sulfonylureas, biguanides, thiazolidinediones, α- glucosidase and glinides as per prescription in Japan.
Arm/Group | Oral Antibiotic Drugs
Number analyzed (Participants) | 162116
Number of Prescriptions
  Dipeptidyl-peptidase 4 inhibitor (DPP4i) | 91634
  Biguanides (BG) | 33238
  Sulfonylurea (SU) | 28211
  α-glucosidase (AGI) | 26192
  Glinide | 16787
  Thiazolidinedione (TZD) | 10344

3. Primary Outcome: Age (Years)
Description: Age of all patients in years calculated for index dates computed from patients in the database. Analysis was done based on index dates used for comparing drugs between the classes. The reported data represent the number of time a prescription was written between 1st January 2014 and 30th September 2016.
Time Frame: From 1st January 2014 to 30th September 2016 (At index date)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Years
Groups:
- Dipeptidyl-peptidase 4 Inhibitor (DPP4i): Patients with type 2 diabetes mellitus (T2DM) were treated with oral antibiotic drug (OAD), Dipeptidyl-peptidase 4 inhibitors (DPP4i), as per prescription in Japan.
- Biguanides (BG): Patients with type 2 diabetes mellitus (T2DM) were treated with oral antibiotic drug (OAD), Biguanide (BG), as per prescription in Japan.
- Sulfonylurea (SU): Patients with type 2 diabetes mellitus (T2DM) were treated with oral antibiotic drug (OAD), Sulfonylureas (SU), as per prescription in Japan.
- α-glucosidase (AGI): Patients with type 2 diabetes mellitus (T2DM) were treated with oral antibiotic drug (OAD), α-glucosidase (AGI), as per prescription in Japan.
- Glinide: Patients with type 2 diabetes mellitus (T2DM) were treated with oral antibiotic drug (OAD), Glinide, as per prescription in Japan.
- Thiazolidinedione (TZD): Patients with type 2 diabetes mellitus (T2DM) were treated with oral antibiotic drug (OAD), Thiazolidinediones (TZD), as per prescription in Japan.
Arm/Group | Dipeptidyl-peptidase 4 Inhibitor (DPP4i) | Biguanides (BG) | Sulfonylurea (SU) | α-glucosidase (AGI) | Glinide | Thiazolidinedione (TZD) | Total
Number analyzed (Participants) | 91634 | 33238 | 28211 | 26192 | 16787 | 10344 | 206406
Years | 71.6 (11) | 66.5 (11) | 72 (11.1) | 71.4 (10.8) | 71.4 (10.8) | 69.7 (11.4) | 70.7 (11.2)

4. Primary Outcome: Sex (Male/Female)
Description: Gender of all patients observed for index dates computed from patients in the database. Results observed were based on index dates used for comparing drugs between the classes. The reported data represent the number of time a prescription was written between 1st January 2014 and 30th September 2016.
Time Frame: From 1st January 2014 to 30th September 2016 (At index date)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Dipeptidyl-peptidase 4 Inhibitor (DPP4i) | Biguanides (BG) | Sulfonylurea (SU) | α-glucosidase (AGI) | Glinide | Thiazolidinedione (TZD) | Total
Number analyzed (Participants) | 91634 | 33238 | 28211 | 26192 | 16787 | 10344 | 206406
Participants
  Female | 36018 | 12681 | 10940 | 9951 | 6549 | 3854 | 79993
  Male | 55616 | 20557 | 17271 | 16241 | 10238 | 6490 | 126413

5. Primary Outcome: Estimated Glomerular Filtration Rate (eGFR)
Description: Estimated glomerular filtration rate (eGFR) was calculated based on the age at index date and the latest serum creatinine at index date (or during the observation period) using formula eGFR millilitre/minute/1.73 meter^2 (mL/min/1.73 m^2) = 194 × (Creatinine)^-1.094 × (age in year)^-0.287 (× 0.739 if female). Analysis was done based on index dates used for comparing drugs between the classes.
Time Frame: Within 6 months from index date
Population: All index dates computed from patients with eGFR data included in the study were considered for this analysis. Some patients were prescribed for more than one study drug and thus we can observe more number of index dates than number of patients.
Measure: Mean (Standard Deviation); unit: millilitre/minute/1.73 meter^2
Arm/Group | Dipeptidyl-peptidase 4 Inhibitor (DPP4i) | Biguanides (BG) | Sulfonylurea (SU) | α-glucosidase (AGI) | Glinide | Thiazolidinedione (TZD) | Total
Number analyzed (Participants) | 11446 | 3523 | 3274 | 3147 | 1890 | 1306 | 25386
millilitre/minute/1.73 meter^2 | 63 (28.8) | 74 (23.9) | 67.4 (26.4) | 60.1 (29.4) | 59.5 (30.2) | 69.7 (23.7) | 65.2 (28.1)

6. Primary Outcome: Prescription Rate of Each Class in Each eGFR Renal Impairment (RI) Level
Description: Renal impairment (RI) is a common complication in patients with type 2 diabetes mellitus (T2DM). Results observed were based on index dates used for comparing drugs between the classes.
Time Frame: Within 6 months from index date
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Dipeptidyl-peptidase 4 Inhibitor (DPP4i) | Biguanides (BG) | Sulfonylurea (SU) | α-glucosidase (AGI) | Glinide | Thiazolidinedione (TZD) | Total
Number analyzed (Participants) | 11446 | 4323 | 3274 | 3147 | 1890 | 1306 | 25386
Participants
  90 < eGFR | 1592 | 838 | 530 | 429 | 252 | 227 | 3868
  60 < eGFR < 90 | 4877 | 2373 | 1446 | 1175 | 691 | 626 | 11188
  30 < eGFR < 60 | 3566 | 1045 | 1090 | 1055 | 610 | 410 | 7776
  eGFR < 30 | 1411 | 67 | 208 | 488 | 337 | 43 | 2554

7. Primary Outcome: Percentage of Concomitant Medications by OAD Classes
Description: Concomitant medication is the drug prescribed other than drug under study in the OAD class on index date. Results observed were based on index dates used for comparing drugs between the classes.
Time Frame: On the index month
Population: as for outcome 2
Measure: Number; unit: Percentage of Prescriptions
Arm/Group | Dipeptidyl-peptidase 4 Inhibitor (DPP4i) | Biguanides (BG) | Sulfonylurea (SU) | α-glucosidase (AGI) | Glinide | Thiazolidinedione (TZD) | Total
Number analyzed (Participants) | 91634 | 33238 | 28211 | 26192 | 16787 | 10344 | 206406
Percentage of Prescriptions
  Use of DPP-4 inhibitors (in %) | 3 | 40 | 32 | 37 | 56 | 34 | 23
  Use of Biguanides (BG) (in %) | 9 | 0 | 11 | 12 | 20 | 19 | 10
  Use of Sulfonylurea (SU) (in %) | 9 | 17 | 1 | 13 | 4 | 21 | 10
  Use of α-glucosidase (AGI) (in %) | 8 | 9 | 6 | 2 | 16 | 10 | 8
  Use of Glinide (in %) | 2 | 3 | 1 | 4 | 4 | 4 | 3
  Use of Thiazolidinedione (TZD) (in %) | 2 | 4 | 2 | 3 | 6 | 1 | 3
  Use of Insulin (in %) | 27 | 23 | 25 | 31 | 37 | 24 | 27

8. Primary Outcome: Percentage of Previous Medications (Premedications) by OAD Classes.
Description: Previous medication is the drug prescribed other than drug under study in the OAD class before index date. Results observed were based on index dates used for comparing drugs between the classes
Time Frame: On the index month
Population: as for outcome 2
Measure: Number; unit: Percentage of Prescriptions
Arm/Group | Dipeptidyl-peptidase 4 Inhibitor (DPP4i) | Biguanides (BG) | Sulfonylurea (SU) | α-glucosidase (AGI) | Glinide | Thiazolidinedione (TZD) | Total
Number analyzed (Participants) | 91634 | 33238 | 28211 | 26192 | 16787 | 10344 | 206406
Percentage of Prescriptions
  Use of DPP4 inhibitors (in %) | 0 | 3 | 2 | 1 | 3 | 8 | 1
  Use of Biguanides (BG) (in %) | 2 | 0 | 1 | 2 | 3 | 2 | 1
  Use of Sulfonylurea (SU) (in %) | 3 | 2 | 0 | 3 | 19 | 2 | 4
  Use of α-glucosidase (AGI) (in %) | 2 | 2 | 1 | 0 | 8 | 1 | 2
  Use of Glinide (in %) | 1 | 1 | 3 | 2 | 0 | 0 | 1
  Use of Thiazolidinedione (TZD) (in %) | 2 | 2 | 1 | 1 | 1 | 0 | 1
  Use of Insulin (in%) | 9 | 7 | 12 | 10 | 12 | 8 | 9

9. Primary Outcome: Percentage of Comorbidities by OAD Classes.
Description: The additional diseases co-occuring, defined by International classification of Diseases, tenth revision (ICD-10) code. Results observed were based on index dates used for comparing drugs between the classes.
Time Frame: On the index month
Population: as for outcome 2
Measure: Number; unit: Percentage of Comorbidities
Arm/Group | Dipeptidyl-peptidase 4 Inhibitor (DPP4i) | Biguanides (BG) | Sulfonylurea (SU) | α-glucosidase (AGI) | Glinide | Thiazolidinedione (TZD) | Total
Number analyzed (Participants) | 91634 | 33238 | 28211 | 26192 | 16787 | 10344 | 206406
Percentage of Comorbidities
  Hypertension (in %) | 69 | 66 | 66 | 70 | 73 | 68 | 68
  Ischemic heart disease (in %) | 30 | 27 | 29 | 33 | 33 | 28 | 30
  Myocardial infarction (in %) | 14 | 13 | 14 | 15 | 14 | 12 | 14
  Heart failure (in %) | 25 | 19 | 23 | 27 | 28 | 19 | 24
  Stroke (in %) | 26 | 22 | 26 | 26 | 27 | 25 | 25
  Renal impairment (in %) | 19 | 10 | 14 | 23 | 26 | 11 | 18
  Diabetic foot (in %) | 9 | 8 | 9 | 10 | 14 | 8 | 9

ADVERSE EVENTS:
Time Frame: Safety reporting is not applicable for this study
Description: The outcomes of the study were the baseline characteristics (pre-treatment) and medication prescriptions. We were not looking at outcomes during the treatment period; therefore safety reporting is not applicable for this study.
Arm/Group | Dipeptidyl-peptidase 4 Inhibitor (DPP4i) | Biguanides (BG) | Sulfonylurea (SU) | α-glucosidase (AGI) | Glinide | Thiazolidinedione (TZD)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The data available was hospital data and not general practitioners data. Only 13.5% patients had laboratory data including eGFR. Some patients who already had other disease compared to the T2DM population were likely to get included in the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-09): https://cdn.clinicaltrials.gov/large-docs/52/NCT03092752/Prot_SAP_000.pdf